CLINICAL TRIAL: NCT02842216
Title: Retrospective Analysis of Hospital Medical Records on Medication and Supplement Use in Pregnant Women
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Michael Ceulemans, PhD Researcher, KU Leuven
Other Study IDs: MC201601
Record Dates: First submitted 2016-07-14; First posted 2016-07-22 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Medication and Supplement Use During Pregnancy
Keywords: Pharmaceutical preparations; Dietary supplements

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Monocentric study in University Hospitals Leuven (campus Gasthuisberg).

Hospital medical records from all pregnant women who delivered between 01/07/2015 and 31/12/2015 in University Hospitals will be analyzed for the presence of medication and supplements.

Some demographic and obstetric parameters will be collected as well.

The anonymized dataset will be analyzed using descriptive statistics (Excel). There will be no intervention among the selected sample.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who delivered in the University Hospital of Leuven between 01/07/2015 and 31/12/2015

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who delivered in the University Hospital of Leuven
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of registered medicines and supplements in hospital medical records of Belgian pregnant women | Hospital medical records from 11 months before delivery until 1 month postpartum

IPD SHARING:
Plan to Share IPD: No